CLINICAL TRIAL: NCT03669939
Title: Toward Safer Opioid Prescribing for Chronic Pain in High Risk Populations: Implementing the Centers for Disease Control Guideline (CDC) Guideline in the Primary Care HIV Clinic.
Brief Title: Toward Safer Opioid Prescribing for Chronic Pain in High Risk Populations
Acronym: TOWER
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The New York Academy of Medicine (Other)
Responsible Party: Principal Investigator, Jessica Robinson-Papp, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-0154
Record Dates: First submitted 2018-08-22; First posted 2018-09-13 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: HIV Disease; Chronic Pain
Keywords: Center for Disease Control Guidelines; Opioids for chronic pain; communication strategies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Chronic Pain | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Communication strategy: Primary Care providers who see HIV patients and follow them on opiates for chronic pain to receive communication strategies developed by the study team wit the guidance from the HV community and providers
  Interventions: Other: Communication Strategy
- Standard of Care: Primary Care Providers - who see HIV patients and follow them on opiates for chronic pain will receive education on the the standard information about the CDC Guidelines
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Communication Strategy — Communication Strategy The intervention consists of a handbook that refers to the CDC Guidelines with tools and communication strategies that the PCP can use when assessing their patients who are on opioids. The Handbook will have a description of the Ohm-app and the information the PCP can retrieve from the dashboard in their medical record. They will also be provided a template to use when seeing the patient to use as guide and as documentation.
  Groups: Communication strategy
Other: Standard of Care — The standard information about the CDC Guidelines and no other information that is available through the study.
  Groups: Standard of Care

SUMMARY:
The overarching plan for TOWER is to develop and test an algorithmic version of the Center for Disease Control Guidelines (CDCG) tailored for a specific primary care setting, the HIV primary care clinic. This CDCG intervention incorporates communication and implementation strategies tailored for the HIV primary care setting, and enabled with technology (an app for use by patients and EMR tools for providers).

DETAILED DESCRIPTION:
However, according to a 2014 AHRQ report, there have been no studies evaluating the effectiveness of any prescription opioid risk mitigation strategies. Furthermore, due to ambiguity in some of the CDCG recommendations and the challenging nature of the patient-provider opioid conversation, the success of the CDCG may hinge on the manner in which it is implemented in individual care settings. Thus it is unclear what the true effect of the CDCG will be. The investigators believe that for the CDCG to have the greatest likelihood of achieving its goals of improving prescription opioid safety without causing unintended effects (e.g. exacerbation of pain, disruption of other aspects of care), its recommendations will need to be skillfully communicated. Furthermore, because of this "human element"and other sources of variability, documenting the effectiveness of the CDCG will require standardization of implementation. The overarching plan for TOWER is to develop and test an algorithmic version of the CDCG tailored for a specific primary care setting, the HIV primary care clinic. This CDCG intervention incorporates communication and implementation strategies tailored for the HIV primary care setting, and enabled with technology (an app for use by patients and EMR tools for providers). Achieving this goal has involved soliciting input from the HIV community using the method of Public Deliberation (PD) in the setting of two Citizen' s Panels, each with ~22 HIV-infected participants and lasting one day; and using the information obtained from the deliberative process to inform the development of the CDCG intervention. The investigators now plan to test the CDCG intervention for feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Attending physician or advance practice provider in one of the Institute of Advanced Medicine (IAM) clinics
* Designated PCP for at least 5 patients to whom he/she prescribes opioids
* Willing and able to adhere to study procedures including randomization, and refraining from discussion of study procedures with other clinical staff or patients

Exclusion Criteria:

* Unwillingness to undergo randomization
* Plans to leave IAM within the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Providers who treat HIV patients in the Institute of Advanced Medicine Institute at Mount Sinai Health System
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible PCPs who successfully complete randomization | 18 months
  Feasibility of recruitment and randomization of PCPs, reflected by the proportion of eligible PCPs who successfully complete randomization (where the denominator is the total number of PCPs offered participation).

SECONDARY OUTCOMES:
Percentage of items in the CDCG intervention which were adhered to | 18 months
  Maintenance of intervention fidelity will be ascertained using the audiotaped data from the clinic visits, and will be described as the percentage of items in the CDCG intervention which were adhered to.

OTHER OUTCOMES:
Standard of Care | 18 months
  Per the CDC guideline (CDCG) for prescribing opioids in general primary care settings, there are 12 recommendations providers must follow in order to reduce prescription opioid-related harms while maintaining pain control and function. In order to monitor providers' adherence to the guideline and to establish appropriateness of "usual care", within the control arm, we will implement the CDCG Adherence Assessment Tool. The CDCG Adherence tool will score patients' EMR notes and will consist of 10-items relevant to the 12 recommendations outlined in the CDCG. If the CDCG recommendations have been denoted in the EMR note, each item will receive points based on a 1-2 numeric scale (max of 16 points). All clinical visits completed during the duration of the study will be scored. A higher number indicating a favorable outcome of adherence to the CDCG guideline.
Primary Outcome Measure determination | 18 months
  The best choice of a primary outcome measure for future studies.
CDCG Adherence Assessment Tool | 18 months
  Two tools will be provided to Intervention providers, an Opioid Managing-app (OM-app) and an EMR note template. The acceptability of the OM-app and EMR tool within the clinical setting will be measured. The OM-app was designed to help collect data needed by the PCP to follow the CDC guideline. The OM-app will contact patients once daily with a link which will take them to a series of questions relevant to their pain management. The app will be responsible for aggregating this data into a report form that the PCP can utilize to facilitate a discussion with the patient and to populate an EMR progress note. The EMR note template will be provided to intervention providers in order to import data collected from the app into a patient's EMR during clinic visits. As with the control arm, the CDCG Adherence Assessment Tool will be implemented which will score patients' EMR notes on a 1-2 numeric scale (max of 16 points). A higher number indicating a favorable outcome.
Current Opioid Misuse Measure (COMM) | 18 months
  17-item, each scored 0 (never) to 4 (very often) with total scale from 0 - 68, higher score indicating more opioid misuse
Self-Reported Misuse, Abuse, and Diversion (SR-MAD) | 18 months
  Self-Reported Misuse, Abuse and Diversion of Prescription Opioids (SR-MAD) instrument consists of 18 self-report items 0-10 numerical rating scale. Total scale from 0 to 180, with higher score indicating worse outcomes.
Brief Pain Inventory (BPI) | 18 months
  Brief Pain Inventory (BPI) is a 9-item instrument with total score from 0 to 10, with higher score indicating worse outcomes.
Hospital Anxiety and Depression Scale (HADS) | 18 months
  14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.
Trust in Provider Scale (TIPS) | 18 months
  11-items scale scored on a 5-point likert scale from 1 (strongly disagree) to 5 (strongly agree). A 52 Freburger et al summary measure of trust is obtained by taking the unweighted mean of the responses to the 11 questions and transforming that value to a 0-100 scale. Higher scores reflect greater trust.
HIV Stigma Scale (HSS) | 18 months
  40-items using a 4 point likert scale 1 (strongly disagree) to 4 (strongly agree), with full scale from 40 to 160. Higher score indicates poorer outcomes
Brief Perceived Ethnic Discrimination Questionnaire-Community Version (BPEDQ-CV) | 18 months
  17-item scale on a summed average likert-type scale from 1 (never happened) to 5 (happened very often). Higher score indicated perception of discrimination.
Internalized Stigma of Chronic Pain (ISCP) | 18 months
  Sum average score on 4-point Likert-type scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Higher score indicates more stigma of chronic pain.
Consumer Assessment of Healthcare Providers and System (CAHPS®) Clinician & Group Survey (CG-CAHPS) | 18 months
  Composite score converted to numerical scale from 0 (never) to 100 (always). and one overall rating of the doctor on a scale from 0 to 10, with higher score showing a more favorable outcome.
Opioid Therapy PROVIDER Survey | 18 months
  10 question survey, sum average score on a 5-point likert scale 1 (strongly agree) to 5 (strongly disagree)
Intervention provider post- survey | 18 months
  6 question survey, intended for provider participants who have been randomized into the intervention arm. The survey includes a 5-point Likert-scale (5=strongly agree, 4=agree, 3=neutral, 2=disagree, 1=strongly disagree) with a high sum average indicating a satisfactory outcome.
Modified ACTG Adherence | 18 months
  A self-reported questionnaire comprised of 8 items. Only item #4 will be used as a percentage of their HIV medication intake, on a scale from 0-100%. . A higher percentage indicating a favorable outcome..
Quantitative Analgesic Questionnaire (QAQ) | 18 months
  Tool for quantifying how much pain meds a patient is taking, by calculating the total weekly doses, the QAQ ("as reported"), and comparing them to the regimen score previously established by physicians who actively treat chronic pain. Regimens are rated on scale from 1 (small amount of meds) to 5 (large amt of meds). 1 QAQ point is assign for taking any opioids at all, & an additional point assign for every equivalent of 100 mg of oral morphine used per week (1-99 mg = 1 pt; 100-199 = 2 pts, etc.). For all other oral meds, 1 point for taking the meds at all, & an additional point for each 25% of the maximum dose taken (1-24% = 1 pt; 25-49% = 2 points, etc.). For topicals, 1 point for each topical reports using regardless of dose or frequency. No upper limit to the amt of QAQ points a patient may accrue. The lowest number of QAQ is 0=no medication. A higher discrepancy between the sum average of QAQ points and "as prescribed" points will indicate a lower adherence rate.
TOWER Post Clinic Visit Interview | 18 months
  This is an 18 item questionnaire of the patients experience after a clinical session with their provider. There are 2 scores, one score will be a sum average on a scale from 0-6 for questions 1-6. The second score will be a sum average on a scale from 0-50 for questions 8-12. A higher scored indicating a favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Robinson-Papp, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical information that is relevant to the provider or patient

REFERENCES:
- [Derived] Cedillo G, George MC, Deshpande R, Benn EKT, Navis A, Nmashie A, Siddiqui A, Mueller BR, Chikamoto Y, Weiss L, Scherer M, Kamler A, Aberg JA, Vickrey BG, Bryan A, Horn B, Starkweather A, Fisher J, Robinson-Papp J. Toward Safer Opioid Prescribing in HIV care (TOWER): a mixed-methods, cluster-randomized trial. Addict Sci Clin Pract. 2022 May 16;17(1):28. doi: 10.1186/s13722-022-00311-8. PMID 35578356